CLINICAL TRIAL: NCT03232775
Title: Evaluating the Effects of a Visual Pedagogy and Structure on the Successful Completion of the Medical Office Visit and Physical Examination With Pre-pubescent Children With Autism
Brief Title: Use of a Visual Pedagogy and Structure With Children With Autism for Routine Physical Exams
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 07-0362
Record Dates: First submitted 2017-07-13; First posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Autism Spectrum Disorder
Keywords: visual pedagogy
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The medical examination teams (one chief medical resident and one nurse) will be blind to the study aim.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Other): Treatment: Physical Exam with Visual Pedagogy and Structure
  Interventions: Other: Treatment: Physical Exam with Visual Pedagogy and Structure
- Control (Other): Control: Physical Exam without Visual Pedagogy and Structure
  Interventions: Other: Control: Physical Exam without Visual Pedagogy and Structure

INTERVENTIONS:
Other: Treatment: Physical Exam with Visual Pedagogy and Structure — Routine physical examination participants receive visual pedagogy and reinforcement (preferred food treat).
  Arms: Treatment
Other: Control: Physical Exam without Visual Pedagogy and Structure — Participants engage in routine physical examination without visual pedagogy and reinforcement (preferred food treat).
  Arms: Control

SUMMARY:
Children with autism spectrum disorders (ASDs) have unique social-communication and behavior impairments that complicate their medical management. This study aimed to evaluate the effectiveness of using a picture schedule paired with a reinforcement system during the medical exam. Two groups (treatment and control) of children (ages 5 - 10 yrs) diagnosed with ASD and below average adaptive communication impairment were asked to participate. Following participation in an overview of autism diagnostic symptoms training, two teams (comprised of one chief medical resident and one nurse), blind to the study aim, conducted the study exams.

DETAILED DESCRIPTION:
Objective: This pilot study aimed to evaluate the effects of a picture-schedule reinforcement system on reducing problem behaviors in children with Autism Spectrum Disorder (ASD) during a physical exam.

Design, setting, patients, intervention: Fifteen study participants, aged 5-10 years, with autism and identified by caregivers as typically uncooperative with physical exams were randomized to one of two physical exam groups (treatment and control) based on their adaptive communication score. The treatment group exam included use of a picture schedule-reinforcement book and the control group exam did not introduce the book. Caregivers rated participants' irritability/stereotypy behaviors before and during study exams. Exam teams blinded to study aims, recorded participants' total exam items completed and caregivers rated participants' level of cooperation.

ELIGIBILITY:
Inclusion Criteria:

1. Chronological ages 4 to 10 years.
2. Presumptive diagnosis of Autistic Disorder or Asperger's Disorder prior to study admission from a psychologist or psychiatrist experienced with children who have autism.
3. Meets research criteria for Autistic Spectrum Disorder:

   1. Meets cut-off scores for autism spectrum on the Social Communication Questionnaire (SCQ) (cut-off = 15) and
   2. Meets empirically-derived algorithm cut-off scores for Autism Spectrum Disorders on the Autism Diagnostic Observation Schedule (ADOS).
   3. All subjects will have the ADOS administered by a clinician trained in research reliability standards.
   4. The Principal Investigator, a certified ADOS trainer and research reliable, or trained designee under the supervision of the Principal Investigator, will administer the ADOS.
4. Participants will represent the typical DSM-IV diagnostic developmental profile of children on the autism spectrum and no neurological injuries or illnesses before the age of three years that could account for their symptoms (i.e., meningitis, encephalitis, severe head injury or seizure disorder).
5. A Communication standard score ≤ 85, as measured by the Vineland Adaptive Behavior Scales - II.

   a) The VABS-II will be administered by the Principal Investigator or trained designee under the supervision of the Principal Investigator as part of the initial phone screening process.
6. Children with an ASD, particularly school-aged children and adolescents, may present with myriad prescribed psychotropic medications. Therefore, we will not exclude children on a variety of psychotropic medications; rather we will conduct a qualitative analysis to look at this issue.
7. No restrictions regarding race or gender will be applied to the autism or developmental disability sample. Every effort will be made not to over-represent any particular race and/or gender group.
8. Physically healthy prior to physical exam.
9. Previous exposure to visual systems. This will be assessed based on caregiver report during the phone screening using one question relating to the use of visual structure with the child.
10. History of:

    1. Poor Cooperation
    2. Completely Uncooperative
    3. Physical exams rated by caregiver on 4-point scale of cooperation modified from Forsberg et al. [56].

       * 0 = No problems with cooperation;
       * 1 = Minor problems with cooperation: Child shows mild behavior problems and/or anxiety symptoms;
       * 2 = Poor cooperation: Child's behavior problems and/or anxiety symptoms requires that the medical staff have to spend extra time and effort to manage the child and complete the exam;
       * 3 = Completely uncooperative: Exam is not possible due to child's behavior problems and/or anxiety symptoms

Exclusion Criteria:

1. Participants with intelligence quotient standard scores > 40.
2. Presence of the following genetic or progressive neurological disorders known to be causative of or potentially resulting in a phenotype similar to autism:

   1. Fragile X,
   2. Landau Kleffner, Rett Disorder,
   3. Childhood Disintegrative Disorder, or
   4. Tuberous Sclerosis, based on screening by clinical staff and subsequent review by medical staff as needed
3. Presence of vision or hearing loss or significant motor impairments.
4. Wards of the State.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline on the Aberrant Behavior Checklist-Community measure ( irritability and stereotypy subscales) | The end of the 15-minute waiting period and within 15 minutes after the completion of physical exam
  Caregiver report form of subjects' behaviors.

SECONDARY OUTCOMES:
Number of study exam items completed during study exams | Within 15 minutes after conclusion of each participant's study exam.
  Study medical personnel teams (nurse and medical resident) tallied number of total exam items completed during study exams with each participant
Change from baseline in Cooperation likert-scale rating form | At study entry and within 15 minutes after the completion of study physical exams
  Caregiver report form of subjects' cooperation behaviors during study physical exams.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Gabriels, PsyD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No